CLINICAL TRIAL: NCT01321203
Title: A Double-blind, Randomized, Controlled Trial of Air Insufflation Versus Carbon Dioxide Insufflation During Endoscopic Retrograde Cholangiopancreatography (ERCP).
Brief Title: Outcome of Carbon Dioxide Versus Air Insufflations During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: DR A. Saravanan Arjunan, Asian Institute of Gastroenterology, India
Other Study IDs: AIG-GI2010-02
Record Dates: First submitted 2011-01-28; First posted 2011-03-23 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Obstructive Jaundice
Keywords: carbon dioxide insufflation
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group-A, use of air;
- Group-B use of CO2

SUMMARY:
To assess the safety and efficacy of CO2 insufflations during ERCP

1. Primary objective:

   To assess the patient's symptoms, abdominal pain and abdominal distension post procedure (ERCP) in the study group.
2. Secondary objective:

Endoscopist:

* To assess the adequacy of bowel distension for adequate luminal visualization
* To assess the peristaltic movement during the ERCP

Anesthetist:

* To measure the PCO2 level in patient post procedure.
* To assess the amount of sedation required during the procedure.
* To assess saturation and vital signs through out the procedure.
* To assess requirement of buscopan.

DETAILED DESCRIPTION:
mentioned in complete

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients referred for ERCP to AIG Hyderabad

Exclusion Criteria:

* Age < 18 years old excluded from the study.
* Patients with COPD.
* Patients with poor ejection fractions and decompensated heart failure.
* Patients with acute illness that require emergency ERCP and not fit for pre procedure and post procedure assessments.
* Patients with recent endoscopic procedure within 24 hours.
* Patient with history of recent surgery within 7 days of duration.
* Pregnant patients.
* Patients not keen to give consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population age group 18yrs and above
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patient comfort post ERCP | 1 hour
  the pain score measures using Visual Analog scale (VAs - 1 to 10 cm scale )

SECONDARY OUTCOMES:
Abdominal distention prior and post ERCP | 5 minutes
  The abdominal girth was measured prior to patient shifted to ERCP table. The immdiately post ERCP the abdominal girth measured. A fixed point is marked at the umblical regiem to maintain the site of abdominal girth.

CONTACTS AND LOCATIONS:
Overall Officials: Saravanan Arjuanan, MD, Principal Investigator — Asian Institute of Gastroenterology, India
Locations (1):
- Asian Institute Of Gastroenterology India, Hyderabad, Andhra Pradesh, India